CLINICAL TRIAL: NCT03064724
Title: Practice-based Intervention for Vietnamese and Korean Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Health Services (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thu Quach, Director of Community Health and Research, Asian Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21BT-0056
Record Dates: First submitted 2017-02-20; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Smoking Cessation; Tobacco Use
Keywords: smoking; tobacco use; Asian; patients; provider advice; digital health intervention
MeSH Terms: conditions — Smoking Cessation; Tobacco Use; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking Cessation Group (Experimental): Patients received the interactive mobile doctor (iMD) intervention.
  Interventions: Behavioral: Interactive Mobile Doctor ("iMD")

INTERVENTIONS:
Behavioral: Interactive Mobile Doctor ("iMD") — iMD delivers tailored interactive video education via a mobile tablet to smoking patients right before their clinic visit with a provider. iMD delivers the "5 A's" (ask, advise, assess, assist, and arrange) and generates a bilingual tailored printout, which aims to increase patient-provider discussion on tobacco use and to promote smoking cessation. This version of iMD delivers the intervention in Korean or Vietnamese languages as preferred by the patient.

SUMMARY:
This pilot project examined the feasibility of an multilingual interactive video education intervention "an interactive Mobile Doctor intervention (iMD)" to promote patient-provider discussion on tobacco use for Korean- and Vietnamese-speaking male patients at primary care settings.

DETAILED DESCRIPTION:
While California has made significant strides in tobacco control and is leading the nation in reducing smoking use, the decline is not observed in all groups. Select groups still have much higher smoking rates and thus bear an unequal burden of tobacco-related illnesses and deaths. Of important note, Asian American men as a combined group have a higher smoking rate than non-Hispanic Whites (22% vs. 18%, respectively); in particular, the highest smoking prevalence has been observed in Vietnamese (31%) and Korean (30%) men among major Asian subgroups. Research also shows that smoking rates are higher for Asian American men with low acculturation (e.g., immigrant status, low English proficiency) than for those who are more acculturated; yet the reverse trend is observed in Asian American women. These findings underscore the need for more targeted tobacco control efforts. The scientific literature suggests that provider advice to quit smoking can influence a smoker's decision to quit. However, research has shown that Asian Americans are less likely to receive such provider advice. Providers often have very limited face-time with patients during the short clinic visit, which presents a challenge as to whether they can incorporate smoking cessation messages during the visit. Overall, little research has focused on smoking cessation in the clinic setting, particularly research that focuses on Asian Americans. The purpose of the pilot study was to develop a more streamlined smoking cessation intervention that can be integrated into the clinic visit, especially to maximize the time when patients are waiting to see their providers. The research question was whether providing culturally appropriate video education that includes provider advice and was tailored to a patient's readiness for quitting smoking will increase whether a patient receives smoking cessation education according to the recommended Clinical Practice Guideline and whether this results in a decrease in tobacco use in low-income Vietnamese and Korean patients. Using a community-based participatory research approach, the investigators created the iMD that delivers tailored in-language video messages via a mobile tablet to Korean and Vietnamese male smokers right before their clinic visit with a provider. iMD delivers the "5 A's" and generates a bilingual tailored printout. Participants were Korean- and Vietnamese-speaking patients who self-identify as daily smokers and receive primary care at a federally-qualified health center. This study evaluated the feasibility and acceptability of iMD from the patients' perspectives. This study examined patient-provider discussion on tobacco use from patients' self-report and electronic health record (EHR), and self-reported quit attempts and smoking abstinence at 3 months post iMD visit.

ELIGIBILITY:
Inclusion Criteria:

* current smokers identified on electronic health records (EHR)
* have a scheduled primary care visit during the recruitment period

Exclusion Criteria:

* already quit smoking or not smoking daily in the past 7 days
* had already quit smoking or not smoking daily in the past 7 days
* had canceled or rescheduled their primary care visit outside of the study period

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Participation Rate | Baseline
  proportion of eligible participants consent to participate
Acceptability | through study completion, an average of 1 year
  proportion of participants who rated the intervention as moderately to extremely satisfied

SECONDARY OUTCOMES:
Patient-provider discussion | "through study completion, an average of 1 year
  self-reported by patient whether discussion on tobacco use took place at the indexed clinical encounter
Physician delivery of 5As | "through study completion, an average of 1 year
  EHR-documented physician's delivery of assess, advice, assist, or arrange at the indexed clinical encounter
Quit attempt | 3-month
  self-reported at least one or more 24 hour quit attempts
Abstinence | 3-month
  self-reported 7-day point prevalent smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Thu Quach, PhD, MPH, Principal Investigator — Asian Health Services; Janice Tsoh, Principal Investigator — University of California, San Francisco